CLINICAL TRIAL: NCT05079529
Title: Development The Potentiality of β-1,3/1,6-D-Glucan (Polysaccharide Peptide) From Mycelia Extract of Indonesia's Ganoderma Lucidum as Adjuvant Therapy in Patients With Cardiometabolic Syndrome Based on NCEP-ATP III Criteria With Modification on Obesity Classification (Waist Circumference Measurement) for Asian Population
Brief Title: Development The Potentiality of β-1,3/1,6-D-Glucan (Polysaccharide Peptide) From Mycelia Extract of Indonesia's Ganoderma Lucidum as Adjuvant Therapy in Patients With Cardiometabolic Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Brawijaya (Other)
Collaborators: PT. Sahabat Lingkungan Hidup (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. dr. Djanggan Sargowo, Sp.PD, Sp.JP(K), Prof, Ph.d, MD, University of Brawijaya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MFBU.DS.PsP021
Record Dates: First submitted 2021-09-18; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Cardiometabolic Syndrome
Keywords: β-1,3/1,6-D-Glucan; Polysaccharide Peptide; Ganoderma lucidum; Cardiometabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: This study conducted cardiometabolic syndrome patients based on NCEP-ATPIII criteria with modification of obesity classification to Asian population criteria. All of the participant would be divided into 2 groups/arms in which one group will be given Polysaccharide Peptide capsule 3 times daily for 90 days and the other one will be given Placebo in the same duration of time.
  Before Polysaccharide Peptide is given, there will be a sequence of pre-test examination, include: blood pressure measurement, body weight and body height measurement to determine Body Mass Index status, waist circumference measurement, blood glucose profile, lipid profile, renal function profile, parameter of inflammation status, parameter of oxidative stress, parameter of endothelial function, and completion of SF 36 questionnaire in which all of them will be done as post-test after intervention completed.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is randomized control double-blinded true experimental study. So the only party that acknowledge whom is given Polysaccharide Peptide capsule or Placebo is the collaborator who provides the adjuvant therapy agent. There is an exception for Outcomes Assessor. They might ask for detail description of the intervention that have been given to the participant if there is any serious adverse event going on.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- β-1,3/1,6-D-Glucan From Mycelia Extract of Indonesia's Ganoderma Lucidum Group (Experimental): This group will receive capsule contains 180 mg of β-1,3/1,6-D-Glucan From Mycelia Extract of Indonesia's Ganoderma lucidum which will be taken 3 times daily for 90 days
  Interventions: Drug: β-1,3/1,6-D-Glucan From Mycelia Extract of Indonesia's Ganoderma Lucidum Group
- Placebo Group (Placebo Comparator): This group will receive empty capsule which will be taken 3 times daily for 90 days
  Interventions: Drug: Placebo Group

INTERVENTIONS:
Drug: β-1,3/1,6-D-Glucan From Mycelia Extract of Indonesia's Ganoderma Lucidum Group — Takes β-1,3/1,6-D-Glucan capsule 3 times daily for 90 days
  Other Names: β-1,3/1,6-D-Glucan
  Arms: β-1,3/1,6-D-Glucan From Mycelia Extract of Indonesia's Ganoderma Lucidum Group
Drug: Placebo Group — Takes placebo capsule 3 times daily for 90 days
  Arms: Placebo Group

SUMMARY:
The aim of this study is to determine the role and efficacy of β-1,3/1,6-D-Glucan (Polysaccharide Peptide) from mycelia extract of Indonesia's Ganoderma lucidum as an antioxidant and anti-inflammatory agent on cardiometabolic syndrome

DETAILED DESCRIPTION:
This study is held at Saiful Anwar General Hospital and General Hospital of Brawijaya University by enrolled 70 participants and using a double-blinded true experimental using a randomized control perspective method with pre-test and post-test design, to determine the effect of giving β-1,3/1,6-D-Glucan (Polysaccharide Peptide) from mycelia extract of Indonesia's Ganoderma lucidum on cardiometabolic syndrome population.

The intended target or experimental variables that will be studied in this study are blood pressure, body mass index, blood glucose profile (fasting glucose, HbA1C), lipid profile (total cholesterol, High-Density Lipoprotein, Low-Density Lipoprotein, and triglyceride), renal function profile (urea and creatinine), heart function from echocardiography examination, inflammation parameter (Interleukin 6, Tumor Necrosis Factor-Alpha, and high sensitivity C-Reactive Protein), stress oxidative parameter (superoxide dismutase and malondialdehyde), endothelial function parameter (nitric oxide), and quality of life that conducted by completion of the SF-36 questionnaire.

Hypothesis of this study is β-1,3/1,6-D-Glucan (Polysaccharide Peptide) from mycelia extract of Indonesia's Ganoderma lucidum can acts as a chronic anti-inflammatory and antioxidant agent in cardiometabolic syndrome patients by contributing in blood pressure control, body mass index control, blood glucose improvement, lipid profile improvement, renal function profile improvement, heart function improvement, and better quality of life. Beside that, the investigators hope that there will be a change of inflammation, stress oxidative, and endothelial function parameter in which shift to the good level.

ELIGIBILITY:
Inclusion Criteria:

* Age more or same than 18 years old
* Defined as metabolic syndrome patients based on NCEP-ATP III Criteria with modified of obesity classification (waist measurement) for Asian population
* Agreed to participate in this study

Exclusion Criteria:

* Allergic to Ganoderma lucidum
* Pregnant woman
* Participate in another drug or medical device study
* Waiting for an organ transplantation or have undergone a transplant
* Cancer patients who undergoing a chemotherapy or radiotherapy
* People with organ failure
* Could not be randomized and participate in this study by clinical judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-12-28 (Estimated); Study Completion 2022-01-06 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life from completion of SF-36 questionnaire | 0 and 90 days
  Quality of Life is assessed by Indonesia validated Short Formm 36 questionnaire. This questionnaire consist of 36 items/questions that evaluate quality of life in some elements. The elements are consisted of changes in health (1 item), general health perception (5 items), energy/fatique (4 items), mental health (5 items), social functioning (2 items), pain (2 items), physical functioning (10 items), role limitations due to emotional problems (3 items) and role limitations due to physical problems (4 items).
  The score from each question will be summed. Minimum score is 36 and maximum score is 138. Higher score indicates higher quality of life and lower score indicates lower quality of life. Higher score after intervention in post-test examination represents a positive outcome

SECONDARY OUTCOMES:
Change of inflammation status parameter (IL-6) level | 0 and 90 days
  Level of IL-6 is obtained from laboratory blood plasma test
Change of inflammation status parameter (TNF-alpha) level | 0 and 90 days
  Level of TNF-alpha is obtained from laboratory blood plasma test
Change of inflammation status parameter (hs-CRP) level | 0 and 90 days
  Level of hs-CRP is obtained from laboratory blood plasma test
Change of oxidative stress parameter (MDA) level | 0 and 90 days
  Level of MDA is obtained from laboratory blood plasma test
Change of oxidative stress parameter (SOD) level | 0 and 90 days
  Level of SOD is obtained from laboratory blood plasma test
Change of endothelial function (NO) parameter level | 0 and 90 days
  Level of NO is obtained from laboratory blood plasma test
Change of waist circumference measurement | 0 and 90 days
  Waist circumference is measured by tape to determine abdominal obesity
Change of body weight and body height measurement | 0 and 90 days
  Body weight is measured by body weight scale and body height is measured by body height scale, then will be combined to determine BMI in kg/m^2
Change of blood pressure | 0 and 90 days
  Blood pressure is measured using manual sphygmomanometer
Change of fasting glucose level | 0 and 90 days
  Fasting glucose level is obtained from laboratory blood test
Change of HbA1C serum level | 0 and 90 days
  HbA1C serum level is obtained from laboratory blood test
Change of triglicyride level status | 0 and 90 days
  Triglyceride level is obtained from laboratory blood test
Change of total cholesterol level status | 0 and 90 days
  Total cholesterol level is obtained from laboratory blood test
Change of HDL level status | 0 and 90 days
  HDL level is obtained from laboratory blood test
Change of LDL level status | 0 and 90 days
  LDL level is obtained from laboratory blood test
Change of creatinine blood level | 0 and 90 days
  Creatinine level is obtained from laboratory blood test
Change of urea blood level | 0 and 90 days
  Urea level is obtained from laboratory blood test

OTHER OUTCOMES:
Number of participants with adverse event (AEs) | 30, 60, and 90 days
  Number of participants that experience adverse event in this study
Number of participants with Serious Adverse Event (SAEs) | 30, 60, and 90 days
  Number of participants that go through serious adverse event in this study

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Brawijaya University (Rumah Sakit Universitas Brawijaya), Malang, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
The research team would like to discuss to what extent and the criteria of individual participant data that will be shared related to Statistical Analysis Plan, Informed Consent Form and/or Clinical Study Report

REFERENCES:
- [Result] Dinh QN, Drummond GR, Sobey CG, Chrissobolis S. Roles of inflammation, oxidative stress, and vascular dysfunction in hypertension. Biomed Res Int. 2014;2014:406960. doi: 10.1155/2014/406960. Epub 2014 Jul 20. PMID 25136585
- [Result] Kharroubi AT, Darwish HM. Diabetes mellitus: The epidemic of the century. World J Diabetes. 2015 Jun 25;6(6):850-67. doi: 10.4239/wjd.v6.i6.850. PMID 26131326
- See also: Journal Title: Vascular Inflammation and Hypertension — https://austinpublishinggroup.com/cardiovascular-diseases/fulltext/ajcd-v3-id1017.php
- See also: Standards of Medical Care in Diabetes — https://www.google.com/url?sa=t&rct=j&q=&esrc=s&source=web&cd=&cad=rja&uact=8&ved=2ahUKEwjt-4mj36_zAhUS5nMBHaFQCYsQFnoECAkQAQ&url=https%3A%2F%2Fcare.diabetesjournals.org%2Fcontent%2Fdiacare%2Fsuppl%2F2016%2F12%2F15%2F40.Supplement_1.DC1%2FDC_40_S1_final.pdf&usg=AOvVaw0Qzl4wVSDwGETFGIa99gJB
- See also: Journal Title: Pathophysiology, Diagnosis and Management of Diabetes Melitus — https://www.google.com/url?sa=t&rct=j&q=&esrc=s&source=web&cd=&cad=rja&uact=8&ved=2ahUKEwjt_eG636_zAhVj5nMBHZexBdkQFnoECAkQAQ&url=https%3A%2F%2Fwww.longdom.org%2Fopen-access%2Fclassification-pathophysiology-diagnosis-and-management-of-diabetesmellitus-2155-6156-1000541.pdf&usg=AOvVaw3TEJc1UhMPP5_lZDYF-Y1z
- See also: Journal Title: Hypertension: Pathophysiology and Treatment — https://www.google.com/url?sa=t&rct=j&q=&esrc=s&source=web&cd=&cad=rja&uact=8&ved=2ahUKEwi5lYHY36_zAhWtuksFHUGjCH8QFnoECAMQAQ&url=https%3A%2F%2Fwww.iomcworld.org%2Fopen-access%2Fhypertension-pathophysiology-and-treatment-2155-9562-5-1000250.pdf&usg=AOvVaw2rNOEbO3b_BS9WrpNQHWVx
- See also: CDC Grand Rounds: A Public Health Approach to Detect and Control Hypertension — https://www.cdc.gov/mmwr/volumes/65/wr/mm6545a3.htm